CLINICAL TRIAL: NCT03949894
Title: Evaluating the Safety and effectivenesS in Adult KorEaN Patients Treated With Tolvaptan for Management of Autosomal domInAnt poLycystic Kidney Disease
Acronym: ESSENTIAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-402-00144
Record Dates: First submitted 2019-04-16; First posted 2019-05-14 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Tolvaptan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tolvaptan (Experimental)
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — 30mg and 15mg of Tolvaptan Tablet
  Other Names: Samsca

SUMMARY:
To evaluate the safety and therapeutic effectiveness of tolvaptan when administered to slow the progression of cyst development and renal function insufficiency in adult Korean patients diagnosed with rapidly progressive ADPKD who have chronic kidney disease (CKD) stages 1-3 at initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily participate by giving written informed consent on this trial
2. Male and female patients aged ≥ 19 to ≤ 50 years
3. Subjects diagnosed with ADPKD based on the Unified Criteria for Ultrasonographic diagnosis of ADPKD (Pei-Ravine Criteria)
4. Subjects with confirmed CKD stages 1-3 at the screening visit
5. Subjects with confirmed rapidly progressive typical ADPKD 'Typical ADPKD'

   * refers to bilateral and diffuse distribution, with mild, moderate or severe replacement of kidney tissue by cysts, where all cysts contribute similarly to TKV.

'rapidly progressive ADPKD'

* Patients will be defined as 'rapidly progressive ADPKD' if they meet any of the following criteria:

  * Mayo class 1C, 1D or 1E

    * Truncating PKD1 mutation confirmed by genetic testing before participating this trial ③ PRO-PKD score > 6 ④ Patients with ADPKD with a decline in Estimated glomerular filtration rate(eGFR) ≥ 5 mL/min/1.73 m2 within 1 year from the screening visit or with an average annual decline in eGFR ≥ 2.5 mL/min/1.73 m2 over a period of 5 years (excluding patients with an eGFR decline due to factors other than ADPKD, such as uncontrolled type 2 diabetes, early diabetic glomerular disease or immune-mediated glomerulonephritis)

Exclusion Criteria:

1. Patients with hyponatremia or hypernatremia
2. Patients with anuria
3. Patients with volume depletion
4. Patients who are unable to sense or appropriately respond to thirst
5. Patients with contraindications to MRI assessment [e.g., ferromagnetic metal prosthesis, aneurysm clips, severe claustrophobia, large tattoo on the abdomen or back, etc.]
6. Patients with severe renal impairment [e.g., patients with currently active glomerulonephritis, kidney cancer, having a single kidney, history of renal surgery within the last 3 years, etc.]
7. Patients with severe hepatic impairment [e.g., cirrhosis, viral hepatitis, unspecified liver function test abnormalities (ALT or Aspartate aminotransferase(AST)) > 3 x ULN or Total Bilirubin > 2 x ULN), etc.]
8. Patients with eGFR decline due to factors other than ADPKD (e.g., uncontrolled type 2 diabetes, early diabetic glomerular disease or immune-mediated glomerulonephritis, etc.)
9. Patients with a history of hypersensitivity and/or specific reactions to benzazepine or benzazepine derivatives (such as Benazepril), or tolvaptan
10. Patients with hereditary problems of galactose intolerance, the Lapp lactose deficiency or glucose-galactose malabsorption, etc.
11. Patients who need chronic diuretic use
12. Patients who are receiving any experimental (not marketed) or approved therapies that may affect the treatment of ADPKD within 6 months from the screening visit [e.g., anti-sense RNA therapy, rapamycin, sirolimus, everolimus and somatostatin analogs (octreotide, sandostatin), vasopressin antagonist (mozavaptan, conivaptan), vasopressin agonist (desmopressin)]
13. Patients who have received cyst decompression or sclerotherapy within 3 years from the screening visit
14. Patients with a history of taking tolvaptan within 6 months from the screening visit
15. Patients who received any investigational medicinal product in another trial within 30 days from the screening visit
16. Fertile women who are currently pregnant or breat feeding, or not willing to use or capable of using acceptable contraceptive methods (abstinence, oral, implanted or injected hormonal methods of contraception, intrauterine device or barrier methods of contraception, such as condom, contraceptive diaphragm and spermicidal agents) to avoid pregnancy until completion of the trial
17. Patients who are, in the opinion of the investigator, unable to comply with the administration of the Investigational Medicinal Product(IMP) or the trial procedures

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
The incidences of TEAEs | during the tolvaptan treatment period and up to 7 days after the date of last dosing
  The incidences of TEAEs
The incidences of TEAEs meeting any of the followings will be summarized. | during the tolvaptan treatment period and up to 7 days after the date of last dosing
  Liver injury [ALT or AST elevation (>3 x ULN) or Total Bilirubin elevation (>2 x ULN), etc.], AEs leading to death, Serious AEs, AEs leading to treatment discontinuation, AEs whose causal relationship with the IMP cannot be ruled out, Severe AEs, Dehydration, Effects on Sodium, Creatinine

SECONDARY OUTCOMES:
Total kidney volume (TKV) annual mean percent change rate [%/year] | from baseline to End of Treatment (Visit 25, Month 24)
  Baseline TKV refers to the value measured during the screening period
eGFR CKD-EPI annual mean change [mL/min/1.73m^2] (off-treatment) | from baseline to the Follow-up visit (Visit 26, 7 days after End of Treatment(Visit 25, Month 24))
  (off-treatment)
eGFR CKD-EPI annual mean change [mL/min/1.73m^2] (on-treatment) | from Completion of Tolvaptan Titration Period (Visit 6, Week 4) to End of Treatment (Visit 25, Month 24)
  (on-treatment)

CONTACTS AND LOCATIONS:
Locations (18):
- South Korea (18):
  - Inje University Busan Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Hallym University Medical Center, Pyeongchon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No